CLINICAL TRIAL: NCT05688202
Title: Simultaneous Versus Sequential Fractional CO2 Laser and Subcision Combination for Post-acne Atrophic Scars: A Split-face Comparative Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ho Chi Minh City Hospital of Dermato-Venereology (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CS/BVDL/22/16
Record Dates: First submitted 2022-12-21; First posted 2023-01-18 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Atrophic Acne Scar
Keywords: Simultaneous; Sequential; Fractional CO2 Laser; Subcision; Combination; Treatment; Split-face; Comparative Study
MeSH Terms: interventions — Lidocaine; Prilocaine; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Each patient will undergo three sessions of subcision combined with fractional CO2 laser with a 1-month interval between sessions. The face's left side is treated with simultaneous combination therapy, in which fractional CO2 laser is performed immediately following subcision. The face's right side receives sequential combination therapy with fractional CO2 laser conducted two weeks after subcision.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left face (Active Comparator): The face's left side is treated with simultaneous combination therapy, in which fractional CO2 laser is performed immediately following subcision
  Interventions: Procedure: Simultaneous combination of fractional CO2 laser and subcision; Device: Fractional CO2 laser; Procedure: Subcision; Drug: Lidocaine/Prilocaine 2.5%-2.5% Topical Application Cream; Drug: Paracetamol; Drug: Lidocaine 2% Injectable Solution
- Right face (Placebo Comparator): The face's right side receives sequential combination therapy with fractional CO2 laser conducted two weeks after subcision.
  Interventions: Procedure: Sequential combination of fractional CO2 laser and subcision; Device: Fractional CO2 laser; Procedure: Subcision; Drug: Lidocaine/Prilocaine 2.5%-2.5% Topical Application Cream; Drug: Paracetamol; Drug: Lidocaine 2% Injectable Solution

INTERVENTIONS:
Procedure: Simultaneous combination of fractional CO2 laser and subcision — Fractional CO2 laser is performed immediately following subcision. Subcision is operated in all participants using an 181/2G Nokor needle (BD Nokor™ Admix Needles, United States). The insertion depth is at the dermal-hypodermal junction. The subcision needle is advanced and retracted in a tunneling motion to penetrate the fibrotic scar tissue, then slid in a direction parallel to the skin's surface in order to detach the scar from its tethers.
  All participants undergo FrCO2 laser (10 600-nm eCO2 laser, Lutronic Corporation, Goyang, Korea) with the parameters following the suggested regimen at static mode: 120 μm beam size, 30 W peak power, 30 - 120 mJ pulse energy, 50-75 spots/cm2 density, with two passes: (1)Only the atrophic scars are treated using a 4mm square or circle pattern, 100-120 mJ pulse energy, and 50 spots/cm2 density. (2)The whole half side of the face is treated using a 12mm square pattern, 30-40 mJ pulse energy, and 75 spots/cm2 density, <10% overlap.
  Arms: Left face
Procedure: Sequential combination of fractional CO2 laser and subcision — Fractional CO2 laser conducted two weeks after subcision. Subcision is operated in all participants using an 181/2G Nokor needle (BD Nokor™ Admix Needles, United States). The insertion depth is at the dermal-hypodermal junction. The subcision needle is advanced and retracted in a tunneling motion to penetrate the fibrotic scar tissue, then slid in a direction parallel to the skin's surface in order to detach the scar from its tethers.
  All participants undergo FrCO2 laser (10 600-nm eCO2 laser, Lutronic Corporation, Goyang, Korea) with the parameters following the suggested regimen at static mode: 120 μm beam size, 30 W peak power, 30 - 120 mJ pulse energy, 50-75 spots/cm2 density, with two passes: (1)Only the atrophic scars are treated using a 4mm square or circle pattern, 100-120 mJ pulse energy, and 50 spots/cm2 density. (2)The whole half side of the face is treated using a 12mm square pattern, 30-40 mJ pulse energy, and 75 spots/cm2 density, <10% overlap.
  Arms: Right face
Device: Fractional CO2 laser — Fractional CO2 laser (10 600-nm eCO2 laser, Lutronic Corporation, Goyang, Korea) on both sides of the face sequentially with a two-week interval between sessions for each face's side by a single physician, with the parameters following the suggested regimen at static mode: 120 μm beam size, 30 W peak power, 30 - 120 mJ pulse energy, 50-75 spots/cm2 density, with two passes. At the first pass, only the atrophic scars are treated using a 4mm square or circle pattern, 100-120 mJ pulse energy, and 50 spots/cm2 density in the static operating mode. At the second pass, the whole half side of the face is treated using a 12mm square pattern, 30-40 mJ pulse energy, and 75 spots/cm2 density in the static operating mode with less than 10% overlap.
Procedure: Subcision — Subcision is operated in all participants using an 1812G Nokor needle (BD Nokor™ Admix Needles, Becton, Dickinson and Company, New Jersey, United States). The operation sites are sterilized with alcohol pads and injected intradermally with a solution of 2% lidocaine. After obtaining appropriate anesthesia, a Nokor needle is inserted into the skin close to the depressed scars and progressed until it lays precisely under the scar. The insertion depth is at the dermal-hypodermal junction. Initially, the subcision needle is advanced and retracted in a tunneling motion to penetrate the fibrotic scar tissue. Once the fibrous mass has been sufficiently fractured, the needle is slid in a direction parallel to the skin's surface in order to detach the scar from its tethers. For densely fibrous scars, several needle insertion sites are used to undermine the defect from various angles.
Drug: Lidocaine/Prilocaine 2.5%-2.5% Topical Application Cream — Preoperative, lidocaine 2.5% and prilocaine 2.5% cream (EMLA 5%, eutectic mixture of local anesthetic; AstraZeneca LP, Wilmington, DE, USA) is applied under occlusion for 60 minutes prior to the removal of local anesthetics
Drug: Paracetamol — A 500 mg paracetamol-based oral analgesic (Efferalgan, Upsa SAS, France) is administered right before the procedure.
  Other Names: Acetaminophen
Drug: Lidocaine 2% Injectable Solution — The operation sites are sterilized with alcohol pads and injected intradermally with a solution of 2% lidocaine.

SUMMARY:
Acne vulgaris, a disease of the pilosebaceous unit, is estimated to afflict 9.4% of the global population, making it the eighth most prevalent and third most significant disease according to the global burden of disease. Post-acne atrophic scars may develop in 95% of acne patients due to aberrant wound healing that affects the pilosebaceous unit and surrounding tissue. Scars are cosmetically unattractive, contributing to the severe psychosocial discomfort observed in acne vulgaris patients.

Several approaches exist for the treatment of post-acne atrophic scars, depending on various factors such as the individual's condition, the types of scars present, and the associated expenses. However, treating atrophic acne scars remains challenging for physicians because there is no gold-standard treatment. Thus, combinations of interventions are typically necessary.

Fractional CO2 laser and subcision are therapeutic methods proven to be effective in treating post-acne atrophic scars. By creating hundreds of thousands of micro-heat treatment zones (MTZs), fractional CO2 lasers emitting small focal spots (50-80 m) via high-focusing mirrors can efficiently treat acne scars. These thermal damage columns accelerate the healing process of collagen synthesis. Subcision, which can be safely paired with other operations, should be the initial step in treating acne scars since it separates scars from underlying structures. Although several studies proposed that the combination of fractional CO2 laser and subcision was more efficacious than a single therapeutic modality, no study has to date compared the efficacy and safety of simultaneous versus sequential combination of these two methods in the treatment of post-acne atrophic scars. There is a critical need for basic research on the effectiveness and adverse events of combining modalities sequentially as compared to simultaneously due to the high expense of traveling and the downtime needed to recover after each treatment, especially for diseases requiring long-term and periodic intervention such as post-acne atrophic scars.

Wound healing is a dynamic process with four distinct but overlapping phases: hemostasis, inflammation, proliferation, and remodeling. The proliferation phase, during which new tissue is formed by a matrix of collagen, elastin, glycosaminoglycans, and other fibrous proteins, begins about four to twenty-one days following an injury. If sequential modalities interfere with each other's proliferative processes, therapeutic efficacy may be compromised. Therefore, our working hypothesis that simultaneous combination is more effective than sequential combination is based on the fact that if the wound-healing process is interrupted, it may stop or progress inadequately. In addition, the investigators anticipate no significant difference between these methods in terms of adverse events frequency and severity, but the downtime in the sequential combination group might be greater than that of the simultaneous combination group. The investigators propose to test the hypothesis by addressing the following two specific aims:

Aim 1: to compare the efficacy and patient satisfaction of simultaneous versus sequential treatment using fractional CO2 laser plus subcision.

Aim 2: To compare adverse reactions of simultaneous and sequential treatment using fractional CO2 laser plus subcision.

Upon completion of this study, the investigators will have (a) compared the treatment outcome of simultaneously versus sequentially combined fractional CO2 laser plus subcision based on ECCA clinical grading score, patient satisfaction, and skin thickness via high-frequency ultrasonography; and (b) compared the incidence and duration of adverse events in simultaneous versus sequential treatment. Optimizing the combination of different interventions will contribute to more efficacious and economical treatment protocols for post-acne atrophic scars.

DETAILED DESCRIPTION:
BACKGROUND

Acne vulgaris and post-acne atrophic scar:

Acne vulgaris, a highly prevalent, multifactorial disorder of the pilosebaceous unit, is characterized by symptomatic discomfort, scarring, emotional and psychological suffering, occupational implications, and the potential for psychiatric disorders, such as depression and suicide. According to the Global Burden of Disease Project, acne has a prevalence of 9.4%, making it the third most significant and the eighth most widespread disease globally.

Post-acne scarring is a permanent, significant consequence of acne vulgaris, affecting 90 to 95 percent of acne patients regardless of severity, with 30 percent suffering from severe scarring. Atrophic scarring is frequently unsatisfactory from an aesthetic standpoint, contributing to the severe emotional distress reported in acne vulgaris patients. One of the primary driving factors for individuals seeking acne treatment is the concern about scarring.

Severity assessment of post-acne atrophic scars is fundamental for patient counseling, appropriate treatment methods selection, treatment efficacy evaluation, and scientific study. Current severity assessment methods of post-acne atrophic scarring involve clinical grading scales such as the ECCA score (echelle d'evaluation clinique des cicatrices d'acne) and objective imaging techniques such as high-frequency ultrasonography.

Treatment of post-acne atrophic scars often involves combinations of modalities since no single treatment method can effectively treat all kinds of scars in every patient. However, the outcome is adversely affected by various factors such as the individual's condition, the types of scars present, the selected treatment methods, and the paradigm of combining these treatment procedures. Until now, there has been no study or consensus in the literature regarding the interval between the two interventions.

Fractional CO2 laser

For more than 20 years, CO2 laser resurfacing has been utilized to treat skin conditions. Initially, they were utilized to cure photoaging, but they are now being used to repair scars caused by trauma, surgery, burns, and acne. Ablative resurfacing involves the use of light-based energy to destroy skin layers. The tissue surrounding the ablative zone is thermally coagulated. After an injury, a reparative mechanism generates new collagen, elastic fibers, and epidermis. Newer versions of CO2 make use of fractionated laser beams as opposed to non-fractionated devices. By doing so, cell columns are preserved, and these untreated ones aid in skin rejuvenation. The development of new collagen and epithelium can improve the appearance of acne scars when applied with fractional lasers. Several advancements have been made in using lasers to treat acne scars over the past several years. The treatment of acne scars has significantly improved by employing combinations of modalities.

Different types of atrophic scars respond inconsistently to fractional CO2 laser. Icepick scars which are narrow and deep to the deep dermis or the hypodermis, respond poorly to fractional CO2 laser. In contrast, rolling scars and shallow boxcar scars can be effectively treated with fractional CO2 laser. Additionally, the treatment effect of fractional CO2 laser is stable and long-lasting, with evidence shown to last until three years after treatment. Common side effects include erythema, swelling, post-inflammatory hyperpigmentation (PIH), pain, crusting, and scaling.

Subcision Orentreich developed subcision in 1995 in order to treat the underlying pathophysiology of rolling acne scars. These scars have a wide, undulating appearance on the skin's surface and lack the clearly defined edges of boxcar and ice pick scars. Rolling scars, despite their superficial appearance, result from deep fibrous attachments connecting the epidermis to the subcutis. Subcision is intended to sever these fibrous bands with minimum harm to the skin's surface. Typically, this procedure raises the depressed scar to the same level as the surrounding skin. David and Norman Orentreich, the inventors of this technology, suggest that the enhancing effect observed following subcision is the product of two separate processes. As soon as the scar base is liberated from its tethers, there is an instantaneous, partial elevation. In the weeks following subcision, it is typical to detect further augmentation of the depressed defect. This following elevation is believed to be the consequence of a wound-healing reaction that culminates in the deposition of new connective tissue beneath the surface of the scar.

Subcision can create long-lasting improvement in the texture of rolling acne scars while inflicting minimal damage to the skin's surface. The technique is simple to perform and typically well tolerated. Despite the possibility of bruising and swelling, the recovery time is short. In addition, the necessary materials are affordable and generally available.

There is no assurance that a single subcision procedure will result in significant improvement. Since the final outcome of the process depends on the individual's unique wound-healing reaction, it is sometimes difficult to anticipate the outcome of the initial therapy. Some individuals require many treatment sessions or additional procedures, like other methods for atrophic scars, such as resurfacing or filler injections, to get optimal results.

Erythema, bruising, edema, and discomfort are typical after subcision and may last for 1-2 weeks. Other uncommon adverse events are the creation of cystic acneiform lesions and hypertrophic or exaggerated responses.

Current paradigms in combining fractional CO2 laser and subcision

Numerous studies have demonstrated that the combination of fractional CO2 laser and subcision is more efficacious than either treatment alone in treating post-acne atrophic scars. In the majority of trials, subcision was done prior to laser treatments, with the interval between the two procedures ranging from simultaneous, one day to two or three weeks. There is a paucity of data concerning the efficacy and safety of therapy combinations with different intervals between procedures. It is unknown whether concurrent operations are more effective than sequential ones. Numerous adverse events of fractional CO2 laser plus subcision have been found in several publications. However, little is known about the differences between the two combination paradigms in terms of side effects.

Hypothesis and aims

Based on current knowledge of the wound healing process and the mechanics of fractional CO2 laser and subcision in treating post-acne atrophic scars, the investigators hypothesize that the simultaneous combination of fractional CO2 laser plus subcision is more efficacious than the sequential combination for the treatment of post-acne atrophic scars. Wound healing is a dynamic process characterized by four distinct but overlapping phases: hemostasis, inflammation, proliferation, and remodeling. The proliferation phase, during which a matrix of collagen, elastin, glycosaminoglycans and other fibrous proteins produce new tissue, begins four to twenty-one days after an injury. If consecutive modalities interfere with each other's proliferative activities, the wound-healing process may be halted or progress insufficiently. In addition, the investigators do not expect a substantial difference between both approaches in terms of the incidence and severity of side effects; however, the downtime in the sequential combination group may be more than that of the simultaneous combination group. The present study is designed to test the above hypothesis by pursuing the following specific aims:

Aim 1: to compare the effectiveness and patient satisfaction of simultaneous versus sequential fractional CO2 laser plus subcision. In this aim, the investigators will conduct a longitudinal study of post-acne atrophic scar patients to identify clinical improvements and patient satisfaction in both treatment groups. Outcomes are assessed via clinical evaluation based on ECCA score and biometrics utilizing HFUS.

Aim 2: to compare the safety of simultaneous versus sequential fractional CO2 laser plus subcision. In this aim, the investigators will utilize the patient population in Aim 1 to identify and compare adverse events in both treatment groups.

Treatment protocol

Each patient will undergo three sessions of subcision combined with fractional CO2 laser with a 1-month interval between sessions. The face's left side is treated with simultaneous combination therapy, in which fractional CO2 laser is performed immediately following subcision. The face's right side receives sequential combination therapy with fractional CO2 laser conducted two weeks after subcision.

Before the procedure

Participants having a history of herpes simplex infection are prescribed oral antiviral tablets containing 400 mg of Acyclovir twice daily for five days, starting two days before the procedure. Preoperative, lidocaine 2.5% and prilocaine 2.5% cream (EMLA, eutectic mixture of local anesthetic; AstraZeneca LP, Wilmington, DE, USA) is applied under occlusion for 60 minutes prior to the removal of local anesthetics. A 500 mg paracetamol-based oral analgesic is administered right before the procedure.

Subcision

Subcision is operated in all participants using an 181/2G Nokor needle (BD Nokor™ Admix Needles, Becton, Dickinson and Company, New Jersey, United States). The operation sites are sterilized with alcohol pads and injected intradermally with a solution of 2% lidocaine. After obtaining appropriate anesthesia, a Nokor needle is inserted into the skin close to the depressed scars and progressed until it lays precisely under the scar. The insertion depth is at the dermal-hypodermal junction. Initially, the subcision needle is advanced and retracted in a tunneling motion to penetrate the fibrotic scar tissue. Once the fibrous mass has been sufficiently fractured, the needle is slid in a direction parallel to the skin's surface in order to detach the scar from its tethers. For densely fibrous scars, several needle insertion sites are used to undermine the defect from various angles.

Laser CO2 fractional

All participants undergo FrCO2 laser (10 600-nm eCO2 laser, Lutronic Corporation, Goyang, Korea) on both sides of the face sequentially with a two-week interval between sessions for each face's side by a single physician, with the parameters following the suggested regimen at static mode: 120 μm beam size, 30 W peak power, 30 - 120 mJ pulse energy, 50-75 spots/cm2 density, with two passes. At the first pass, only the atrophic scars are treated using a 4mm square or circle pattern, 100-120 mJ pulse energy, and 50 spots/cm2 density in the static operating mode. At the second pass, the whole half side of the face is treated using a 12mm square pattern, 30-40 mJ pulse energy, and 75 spots/cm2 density in the static operating mode with less than 10% overlap.

After the procedure

Right after the procedure, participants' faces are cooled by wet dressings with NaCl 0.9%, and sterilized gauze is applied to cover the treated area. Following subcision, antibiotic ointment and oral antibiotics may be prescribed.

Statistical method

Statistical analyses are performed using R 4.2.2 binary for macOS (Big Sur), Apple silicon Macs (M1). Continuous variables with normal distributions are presented as mean (standard deviation) and median (minimum-maximum) for those with abnormal distributions. Categorial variables are summarized as frequencies and percentages. Student's t-test or Mann-Whitney-Wilcoxon test are used to show the differences between dependent numerical groups with and without normal distribution, respectively. Paired t-test or Wilcoxon Signed Rank is used to compare continuous variables in the same group. For dichotomous variables, the Chi-squared test or Fisher is used as appropriate. A p-value less than 0.05 is considered significant.

INNOVATION AND CREATIVITY STATEMENT

Post-acne atrophic scars treatment, either single or combined intervention, poses a major challenge for physicians. More importantly, prolonged downtime and irritated adverse events prevent patients from adhering long time treatment. This project and its methodology represent an essential shift in the strategy of combining different methods for treating post-acne atrophic scars, thereby contributing to better treatment and reducing adverse events.

A clarification in paradigm

Currently, there are two approaches of combination between fractional CO2 laser and subcision: sequential combination (in which two interventions are performed days to weeks apart) and simultaneous combination. Each of these strategies has major disadvantages. The sequential treatment downtime is prolonged, and its adherence is poor since patients must pay multiple time-consuming visits to pursue it. Because simultaneous treatment is assumed to associate with more severe skin damage and side effects such as pain and swelling, simultaneous combination remains limited in routine clinical practice. Until now, there has been no study or consensus on the interval between the two interventions.

Our project represents a radical clarification of the current paradigm. By comparing the efficacy and safety of different combination strategies, the investigators can identify a better combination method to effectively treat post-acne atrophic scars.

Advanced method for objective assessment

Apart from treatment evaluation using clinical score scales (ECCA score) based on photographs, our project assesses treatment efficacy by measuring biometrics utilizing high-frequency ultrasonography.

So far, the majority of publications have utilized photographs and interviewed patients receiving treatment about their satisfaction with therapeutic effects to evaluate acne scars and treatment outcomes. This approach gives a preliminary assessment of the treatment, although it is subjective and lacks precision. There have been a few reports of histologic research, but they are invasive. This diagnostic gap may be filled by high-frequency ultrasonography (HFUS). It has been used in dermatology for more than 20 years to study and quantify skin changes associated with various diseases. This imaging technology enables precise measurements of skin thickness. It has been demonstrated that HFUS is objective, reliable, and safe for the patient in several fields of dermatology, cosmetology, and aesthetic medicine.

SIGNIFICANT STATEMENT

Our project has clinical significance as it will address an unmet need and allow an improved treatment paradigm with more efficacy, safety, and convenience.

Addressing an unmet clinical need

Acne vulgaris is the third most burden disease, and post-acne atrophic scars inflict more than 95% of acne patients. Despite recent progress in treatment, post-acne atrophic scar patients still have poor outcomes. There are multiple methods for treating post-acne atrophic scars based on considerations such as the individual's condition, the scar types present, and the associated expenditures. However, treating atrophic acne scars remains difficult because there is no best therapy for this condition. Consequently, combinations of interventions are becoming a new essential trend and are more widely used. These practical needs have raised questions about the combination paradigm's aspects, such as interventional timing, efficacy, and safety.

Improving treatment paradigm

Efficacy and safety present major challenges to the treatment of post-acne atrophic scar patients since clinical improvements require multiple treatment sessions and a long follow-up time to observe. Moreover, side effects often occur and take extended downtime to recover, which are irritable or unacceptable to some patients. However, improvements in scar appearance are sometimes modest. As interventional timing plays an essential role in combining different therapeutic modalities, comparing simultaneous and sequential combinations helps physicians to select a more effective therapeutic paradigm and hence improve treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post-acne atrophic scars on both facial sides visiting HCMC Hospital of Venereology and Dermatology in the conducting period;
* Agreement to give written informed consent and authorization for release of personal health data.

Exclusion Criteria:

* Patients in pregnancy or lactation
* Patients who use oral isotretinoin within the preceding six months or topical retinoids (tretinoin, retinol, tazoretin, tazarotene) within the preceding two weeks
* Patients with active moderate-severe acne vulgaris
* Patients with a history of keloid/hypertrophic scar formation
* Patients undergone cosmetic procedure (filler injections, botulinum toxin A, ablative/non-ablative laser resurfacing procedures, chemical reconstruction of skin scars, collagen induction therapy using a microneedle therapy system at the treatment site within the preceding six months
* Patients undergoing immunosuppressive therapy
* Patients currently using anticoagulative or antiplatelet medications
* Patients with active infections at the treatment sites; (i) patients with systemic diseases (heart failure, diabetes,…)
* Patients with active Herpes simplex infections at the treatment sites.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline skin thickness at 3 months after the last treatment session. | Change from baseline and 3 months after the last treatment session
  Before the treatment and three months after the final session, a high-frequency ultrasound system (Supersonic Mach 30, Hologic, SuperSonic Imagine, Aix-en-Provence, France), which uses a 20 MHz linear probe with 8mm penetration, 30x12m um resolution, provides a quantitative assessment and measurements in mm. Acquired HFUS images are imported into MATLAB's image segmenter to segment and delineate skin layers. A MATLAB code is applied to assess skin thickness from segmented images. The skin's overall thickness, epidermis, and dermis at the treatment sites are also measured (unit: mm).
Change from baseline skin thickness at 6 months after the last treatment session. | Change from baseline and 6 months after the last treatment session
  Before the treatment and six months after the final session, a high-frequency ultrasound system (Supersonic Mach 30, Hologic, SuperSonic Imagine, Aix-en-Provence, France), which uses a 20 MHz linear probe with 8mm penetration, 30x12m um resolution, provides a quantitative assessment and measurements in mm. Acquired HFUS images are imported into MATLAB's image segmenter to segment and delineate skin layers. A MATLAB code is applied to assess skin thickness from segmented images. The skin's overall thickness, epidermis, and dermis at the treatment sites are also measured (unit: mm).
ECCA score at baseline | Baseline
  The ECCA score (echelle d'evaluation clinique des cicatrices d'acne) provides a quantitative grading score for evaluating scars' severity and clinical improvement, with a minimum - maximum value is 0 - 540. A higher score means higher severity of acne scars condition.
ECCA score at week 4 | Week 4
  The ECCA score (echelle d'evaluation clinique des cicatrices d'acne) provides a quantitative grading score for evaluating scars' severity and clinical improvement, with a minimum - maximum value is 0 - 540. A higher score means higher severity of acne scars condition.
ECCA score at week 8 | Week 8
  The ECCA score (echelle d'evaluation clinique des cicatrices d'acne) provides a quantitative grading score for evaluating scars' severity and clinical improvement, with a minimum - maximum value is 0 - 540. A higher score means higher severity of acne scars condition.
ECCA score at Week 12 | Week 12
  The ECCA score (echelle d'evaluation clinique des cicatrices d'acne) provides a quantitative grading score for evaluating scars' severity and clinical improvement, with a minimum - maximum value is 0 - 540. A higher score means higher severity of acne scars condition.
ECCA score at 3 months after the last treatment session. | 3 months after the last treatment session.
  The ECCA score (echelle d'evaluation clinique des cicatrices d'acne) provides a quantitative grading score for evaluating scars' severity and clinical improvement, with a minimum - maximum value is 0 - 540. A higher score means higher severity of acne scars condition.
ECCA score at 6 months after the last treatment session. | 6 months after the last treatment session.
  The ECCA score (echelle d'evaluation clinique des cicatrices d'acne) provides a quantitative grading score for evaluating scars' severity and clinical improvement, with a minimum - maximum value is 0 - 540. A higher score means higher severity of acne scars condition.
Investigator's Global Assessment at Week 4 | 4 weeks after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by a blinded investigator is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Investigator's Global Assessment at Week 8 | 8 weeks after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by a blinded investigator is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Investigator's Global Assessment at Week 12 | 12 weeks after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by a blinded investigator is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Investigator's Global Assessment at 3 months | 3 months after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by a blinded investigator is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Investigator's Global Assessment at 6 months | 6 months after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by a blinded investigator is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Patient's Global Assessment at Week 4 | 4 weeks after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by patients is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Patient's Global Assessment at Week 8 | 8 weeks after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by patients is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Patient's Global Assessment at Week 12 | 12 weeks after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by patients is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Patient's Global Assessment at 3 months | 3 months after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by patients is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Patient's Global Assessment at 6 months | 6 months after the last treatment session.
  Photographs (five photos taken at 0,45 and 90 degrees of each half face, and multiple close-ups at the scar sites) are taken at baseline, before each treatment session, and three months after the last session. When comparing images taken prior to and after therapy, the head's position, distance from the camera, and illumination remain constant. Evaluation of global assessment to treatment by patients is done using patient photographs of before and after treatment. Rating the Investigator's Global Response to treatment is done using a quartile grading scale (0 = no improvement 0%; 1 = mild improvement 1% - 25%;2 = moderate improvement 25%-49%; 3 = significant improvement 50%-74%; 4= marked improvement ≥ 75%).
Patients Satisfaction | 6 months after the last treatment session.
  Patients are asked to rate their satisfaction with each type of combination therapy on a four-point Likert scale with the following anchors: extremely satisfied, satisfied, partially satisfied, and dissatisfied.

SECONDARY OUTCOMES:
Pain level after laser | Baseline (right after first treatment session)
  Pain level is documented (using a ten-point Visual Analog Scale). Patients will be asked to rate their pain level on the scale of 10 (minumum: 0, no pain; maximum: 10, extremely pain)
Pain level after laser | Week 4 (right after second treatment session)
  Pain level is documented (using a ten-point Visual Analog Scale). Patients will be asked to rate their pain level on the scale of 10 (minumum: 0, no pain; maximum: 10, extremely pain)
Pain level after laser | Week 8 (right after third treatment session)
  Pain level is documented (using a ten-point Visual Analog Scale). Patients will be asked to rate their pain level on the scale of 10 (minumum: 0, no pain; maximum: 10, extremely pain)
Pain level after subcision | Baseline (right after first treatment session)
  Pain level is documented (using a ten-point Visual Analog Scale). Patients will be asked to rate their pain level on the scale of 10 (minumum: 0, no pain; maximum: 10, extremely pain)
Pain level after subcision | Week 4 (right after second treatment session)
  Pain level is documented (using a ten-point Visual Analog Scale). Patients will be asked to rate their pain level on the scale of 10 (minumum: 0, no pain; maximum: 10, extremely pain)
Pain level after subcision | Week 8 (right after third treatment session)
  Pain level is documented (using a ten-point Visual Analog Scale). Patients will be asked to rate their pain level on the scale of 10 (minumum: 0, no pain; maximum: 10, extremely pain)
Other adverse events | Week 4
  Other adverse effects are also documented (Yes or No) including post-inflammatory hyperpigmentation, post-inflammatory hypopigmentation, and other side effects using a questionnaire assessing adverse events.
Other adverse events | Week 8
  Other adverse effects are also documented (Yes or No) including post-inflammatory hyperpigmentation, post-inflammatory hypopigmentation, and other side effects using a questionnaire assessing adverse events.
Other adverse events | Week 12
  Other adverse effects are also documented (Yes or No) including post-inflammatory hyperpigmentation, post-inflammatory hypopigmentation, and other side effects using a questionnaire assessing adverse events.
Erythema | Week 4
  The duration (unit: days) of erythema presented after a treatment session
Erythema | Week 8
  The duration (unit: days) of erythema presented after a treatment session
Erythema | Week 12
  The duration (unit: days) of erythema presented after a treatment session
Edema | Week 4
  The duration (unit: days) of edema presented after a treatment session
Edema | Week 8
  The duration (unit: days) of edema presented after a treatment session
Edema | Week 12
  The duration (unit: days) of edema presented after a treatment session
Crusting | Week 4
  The duration (unit: days) of crusting presented after a treatment session
Crusting | Week 8
  The duration (unit: days) of crusting presented after a treatment session
Crusting | Week 12
  The duration (unit: days) of crusting presented after a treatment session
Bruising | Week 4
  The duration (unit: days) of bruising presented after a treatment session
Bruising | Week 8
  The duration (unit: days) of bruising presented after a treatment session
Bruising | Week 12
  The duration (unit: days) of bruising presented after a treatment session
Downtime | Week 4
  Total downtime duration (unit: days) needed for recovery after a treatment session
Downtime | Week 8
  Total downtime duration (unit: days) needed for recovery after a treatment session
Downtime | Week 12
  Total downtime duration (unit: days) needed for recovery after a treatment session
Lump | 3 months after last treatment session
  The duration of lump presented after 3 treatment sessions (Ordinal variable with 7 values: 0 - no lump; 1 - 1 month; 2 - 2 months; 3 - 3 months; 4 - 4 months; 5 - 5 months; 6 - > 5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Quoc Bao Tran, Doctor, Principal Investigator — Ho Chi Minh City Hospital of Dermato-Venereology
Locations (1):
- Ho Chi Minh City Hospital of Dermato - Venereology, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded and updated to datadryad.org
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Information of request reviewer:
  Name: QUOC BAO TRAN Phone number: (+84) 934181096 Email: baotran181019996@gmail.com Address: 02 Nguyen Thong, Ward Vo Thi Sau, District 3, Ho Chi Minh City, Vietnam